CLINICAL TRIAL: NCT01951092
Title: mHealth Intervention Supporting HIV Treatment Adherence and Retention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Miriam Hospital (Other)
Responsible Party: Principal Investigator, Aadia Rana, Assistant Professor of Medicine, The Miriam Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Lifespan Dev Grant Rana-2012
Record Dates: First submitted 2013-09-18; First posted 2013-09-26 (Estimated); Results first posted 2016-04-22 (Estimated); Last update posted 2016-04-22 (Estimated); Status verified 2016-04

CONDITIONS: HIV; Adherence; Retention
Keywords: HIV; adherence; retention; texting

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single Arm intervention study (Experimental): All subjects receive text messages for: 1) medication reminders; 2) appointment reminders; 3) a text message addressing barriers (e.g., reminders to attend AA meetings). Each subject will undergo baseline assessments, choose personalized messages at that time. Subsequently monthly phone calls with study coordinator regarding frequency/changing messages, and then month 3 assessment, and month 6 (final assessment) with option for qualitative interview.
  Interventions: Other: Text messaging

INTERVENTIONS:
Other: Text messaging

SUMMARY:
Despite advances in antiretroviral treatment (ART) over the past 10 years, the incidence of HIV in the United States remains stagnant with over 50,000 new cases annually. HIV-infected individuals inconsistently engaged with care are less likely to receive ART which is associated with correspondingly adverse clinical outcomes in the long term and increased risk of transmission. Mobile health (mHealth) strategies including cell phone and text messaging have shown success in the developing world for medication adherence, yet mHealth interventions have not been developed to improve retention in HIV care. This strategy needs to be tested to demonstrate feasibility, acceptability and preliminary effectiveness in supporting HIV treatment adherence in Rhode Island.

The Miriam Hospital Immunology Center is an urban HIV-clinic that provides comprehensive primary and specialty care for over 1400 HIV-infected patients. It is the largest HIV clinic in Rhode Island with patients also referred from eastern Connecticut and southern Massachusetts. In 2010, there were 165 new patients in clinic, 70 of whom were diagnosed within 1 year of entering care. In this environment, we propose a pilot study with the following specific aims:

Specific Aim 1: To pilot a bidirectional mHealth intervention among individuals at high risk of loss to follow-up, including those with a recent HIV diagnosis or those re-engaging in HIV care. HIV-infected persons (n=30) with a recent diagnosis or re-engaging in care at the Immunology Center at TMH will be recruited to participate in a bidirectional mHealth intervention that delivers automated, regularly scheduled appointment and medication adherence reminders in an individualized format, and also allows individuals to request motivational enhancement and problem-solving support to address barriers to care.

Specific Aim 2: To assess the impact and acceptability of the pilot intervention through qualitative interviews. All participants will also be invited to complete individual in-depth interviews which will assess acceptability and effectiveness of the pilot mHealth intervention, such as content and frequency of automatic messages, for retention and medication adherence for HIV-infected individuals in RI.

The results of this study will provide preliminary data to inform an R21 or R34 application to determine efficacy of an mHealth intervention among HIV-infected persons at high-risk for loss to follow-up.

ELIGIBILITY:
Inclusion Criteria:

* HIV infected
* age >/= 18
* patient at The Miriam Hospital Immunology Center
* has cell phone that can send and receive text messages
* English speaking only

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2013-02; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- The Miriam Hospital Immunology Center, Providence, Rhode Island, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients at the Immunology Center in Providence RI who were either 1) newly diagnosed, 2) returning to care after a gap, 3) or with difficulties with adherence to care were eligible for enrollment in this pilot study.
  Participants were recruited from January 2013 through July 2013 and followed for 6 months.
Groups:
- Single Arm Intervention Study: All subjects receive text messages for: 1) medication reminders; 2) appointment reminders; 3) a text message addressing barriers (e.g., reminders to attend AA meetings). Each subject will undergo baseline assessments, choose personalized messages at that time. Subsequently monthly phone calls with study coordinator regarding frequency/changing messages, and then month 3 assessment, and month 6 (final assessment) with option for qualitative interview.
  Text messaging
Period: Overall Study
Arm/Group | Single Arm Intervention Study
Started | 32
Completed | 20
Not Completed | 12
Not completed — Lost to Follow-up | 10
Not completed — Incarceration | 1
Not completed — Transfer of Care | 1

BASELINE CHARACTERISTICS:
Arm/Group | Single Arm Intervention Study
Number analyzed (Participants) | 32
Age, Continuous [Median (Full Range); unit: years] | 36 [19 to 64]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 22
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 20
  More than one race | 2
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 32
Participants with HIV PVL <200 copies/mL [Number; unit: participants] — Number of patients with baseline HIV PVL <200 copies/mL
  participants | 18

OUTCOME MEASURES:

1. Primary Outcome: Number of Particpatns Who Considered the Intervention Feasible and Acceptable
Description: A qualitative interview is completed at the end of the 6 month intervention where participants are queried on aspects of the texting intervention including: frequency of messaging, content of messaging, comfort with confidentiality with messaging, interactions between clinic staff as a result of messaging, and ideas on how to incorporate messaging clinic-wide.
Time Frame: 6 months
Population: All 20 participants who completed the study at 6 months participated in interviews and reported that the texting intervention was feasible and acceptable.
Measure: Number; unit: participants
Arm/Group | Single Arm Intervention Study
Number analyzed (Participants) | 20
participants | 20

2. Secondary Outcome: Efficacy
Description: Exploratory end point of PVL <200 copies at the end of the study
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | Single Arm Intervention Study
Number analyzed (Participants) | 32
participants | 32

ADVERSE EVENTS:
Time Frame: 6 months (during participation in the study)
Description: Primary adverse events evaluated for would be loss of confidentiality due to text messaging. None were reported in this study.
Arm/Group | Single Arm Intervention Study
Serious Adverse Events (participants affected / at risk) | 0/32
Other Adverse Events (participants affected / at risk) | 0/32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No